CLINICAL TRIAL: NCT02510508
Title: A Group Version of Community Reinforcement and Family Training (CRAFT) Compared to Self-Directed CRAFT Delivery and Non-intervention: a Three-armed Randomized Clinical Trial
Brief Title: Group Version of CRAFT Compared to Self-Directed CRAFT Delivery and Non-intervention: a Three-armed RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants were included
Sponsor: IrisZorg (Other)
Responsible Party: Principal Investigator, Hendrik Roozen, Ph.D, IrisZorg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL48307.028.14
Record Dates: First submitted 2015-07-16; First posted 2015-07-29 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Addiction; Substance Use Disorder; Alcohol Use Disorder; Substance- Related Disorder
Keywords: addiction; substance abuse; alcohol; drugs; community reinforcement; family treatment; randomized control trial
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group CRAFT (Experimental): All CSO's who are allocated to CRAFT group condition will be offered seven sessions of a CRAFT Group format. Each group will meet for 90 minutes weekly and will be completed within 2 months. The group content is based on the CRAFT techniques described by a training manual written by Roozen, Smith and Meyers (2015). Furthermore the CSOs in this condition will also receive a Dutch version of the CRAFT self-help book (Self Directed CRAFT Delivery), "Get your loved one sober: Alternatives to nagging, pleading and threatening" (Meyers & Wolfe, 2012). Groups will engage in a combination of didactic teaching, role-play of new communication styles and discuss their experiences utilizing CRAFT skills.
  Interventions: Behavioral: Group CRAFT; Other: Non-intervention
- Self-Directed CRAFT Delivery (Active Comparator): CSO's allocated to the Self- Directed CRAFT Delivery will receive the Dutch version of the CRAFT self-help book, "Get your loved one sober: Alternatives to nagging, pleading and threatening" (Meyers & Wolfe, 2012). The book helps CSO's how to utilize the CRAFT model in their daily lives. It includes guidelines for responding to IP behavior, improving positive communication skills, improving the CSO's own well-being and explains how to engage the IP into treatment.
  Interventions: Behavioral: Self-Directed CRAFT Delivery; Other: Non-intervention
- Non-intervention (No Intervention): Participants assigned to the non-intervention condition will be placed on a Group CRAFT waiting list.

INTERVENTIONS:
Behavioral: Group CRAFT — CSOs will receive seven weekly 90 min sessions of CRAFT + Self-Directed CRAFT Delivery
  Arms: Group CRAFT
Behavioral: Self-Directed CRAFT Delivery — CRAFT self-help book (Self Directed CRAFT Delivery)
  Other Names: CRAFT self-help book condition
  Arms: Self-Directed CRAFT Delivery
Other: Non-intervention — Non-intervention
  Other Names: Waitinglist condition
  Arms: Group CRAFT; Self-Directed CRAFT Delivery

SUMMARY:
The aim of this study is to determine whether a group format Community Reinforcement and Family Training (CRAFT) and Self-Directed CRAFT Delivery are more effective than non-intervention in terms of Concerned Significant Others (CSO) well- being and cost- effectiveness.

DETAILED DESCRIPTION:
The aim of this study is to determine the applicability and effectiveness of (a) CRAFT group format in conjunction with the CRAFT self-help book and (b) a CRAFT self-help book (self-directed CRAFT delivery condition), compared to (c) non-intervention (control). The primary aim is increase CSO well- being and reduce CSO health complaints. CSOs will be assessed at baseline (T0), 2 months (end of intervention) (T1), 3 months- (T2), and 6 months follow-up (T3), independently of the assigned condition. Secondary outcomes will encompass cost-effectiveness of both CRAFT interventions. Also, we measure IP engagement and IPs' substance use.

Since the negative consequences of substance abuse are not limited to alcohol- and drug users themselves, it also affects the lives of family members and close friends (CSOs). This study focusses on CSOs to improve their lives. Recruitment will take place in the Netherlands (nation- wide). Assessment and the CRAFT group intervention will be conducted at six different locations (Arnhem, Doetinchem, Ede, Nijmegen, Tiel and Zevenaar, all in the province of Gelderland) in the Netherlands. Participants will be recruited via advertisements on the Internet, social media, websites of IrisZorg (centre for addiction care and sheltered housing ), and subsequently, in local newspapers and flyers located in emergency rooms, general practitioners, family practice clinics, and mental health based treatment agencies.

To obtain information about the presence of psychiatric disorders of the CSOs, a Dutch version of the Mini-International Neuropsychiatric Interview (M.I.N.I.) will be used. After initial assessment, a randomization procedure will be conducted by an independent researcher, who is affiliated to the Erasmus Medical Center, Rotterdam, the Netherlands. CSOs will be informed about the allocation of conditions within 1 week, after initial admission. Several outcome measures will be used in this study. The following will be measured:

1. CSO well- being (including physical and psychological health and complaints, quality of life, quality of the relationship, self- efficacy and social support);
2. cost-effectiveness of both CRAFT and Self- Directed Delivery compared to non- intervention.
3. IP engagement and IP substance use.

Using the primary outcome, CSO well-being, a priori power analysis is completed. Means and standard deviations for CSO well-being, measured with the Beck Depression Inventory (BDI), for Group CRAFT were used (Miller et al., 1999). An effect size was calculated (f = 0.22). The power analysis, conducted with the online program called G-power, indicated that a total sample size of 69 CSOs is needed to achieve a power of 95% for detecting a medium effect size when using the p = 0.05 criterion of statistical significance. These numbers are based on an ANOVA with a within-between subject design. Based on the pilot study of Kirby et al. (1999), 23% drop out after 3- and 6- month follow-up is taken into account. This means that, including the 23% drop-out-rate and based on the sample size of 69, an N of 85 is needed after 3 months and that a total N of 105 is needed to complete all assessments. Summarized, to be able to have at least 69 assessments completed at 6- month follow- up, a total sample size of 105 CSOs is required; with an estimated total drop-out rate of 34%.

ELIGIBILITY:
Inclusion Criteria:

* CSO has concern about and having direct knowledge of alcohol- and/or drug problems of an IP, who is either a first degree relative, intimate partner or close friend.
* Age at least 18 years (the CSO)
* Reports that IP is not currently in addiction treatment (at IrisZorg and elsewhere) and has not received addiction treatment in the past 3 months
* Reports that IP is treatment-refusing
* Evidence (according CSO) that the IP meets criteria for SUDs according to The Structured Clinical Interview for DSM IV axis 1 Disorders (SCID-I)

Exclusion Criteria:

* Does not demonstrate an adequate understanding of their participation, informed consent, and requirements of the protocol, or has insufficient reading abilities to comprehend the Dutch self-help book or does not agree to participate by refusing to sign an informed consent
* CSO meets the DSM-IV criteria for any current SUD diagnosis, through clinical assessment by The Structured Clinical Interview for DSM IV axis 1 Disorders (SCID-I) and the Dutch version of the Mini- International Neuropsychiatric Interview ( M.I.N.I.)
* Refuses to provide valid locator information, allow audiotaped sessions, and/or participate in follow-ups
* Evidence that the IP had received treatment (other than detoxification) for alcohol or drug problems in the prior three months, was mandated by the courts to receive treatment, or was currently motivated to accept treatment
* IP has a recent history of severe domestic violence
* CSO is involved in a concomitant intervention to get the IP in treatment or to improve their own well-being
* CSO fails to complete less than 4 Group CRAFT sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Concerned Significant Other (CSO) well-being (physical and psychological) | 4 months after the initiation of the intervention
  Measured by the following tests:Measurement of the Addictions for Triage and Evaluation (MATE), Depression Anxiety Scales (DASS-21), Maudsley Addiction Profile (MAP), Research and Development- 36 (RAND- 36), Trimbos/iMTA questionnaire for Costs Associated with Psychiatric Illness (TicP) and EuroQol- 5D.

SECONDARY OUTCOMES:
CSO quality of life | 4 months after the initiation of the intervention
  Measured by the following tests: CRA- Happiness Scale (CRA-HS) and WHOQol- Bref
CSO quality of the relationship | 4 months after the initiation of the intervention
  Measured by the following tests: CRA Relationship Happiness Scale (CRA-RHS), Agression Questionnaire (AQ) and Experiences in Close Relationships Scale- short form (ECR)
Other CSO reported psychological measures | 4 months after the initiation of the intervention
  Measured by the following tests: General Self-Efficacy Scale (GSES) and Social Support Inventory (SSI).
Cost-effectiveness of group CRAFT and Self-Directed CRAFT Delivery compared to non-intervention condition | 4 months after the initiation of the intervention
  Measured by: TiC-P; EuroQol- 5D and RAND-36

OTHER OUTCOMES:
Identified Patient (IP) engagement for all three conditions | 4 months after the initiation of the intervention
  Attending at least 1 treatment session
CSO Drop-out | 4 months after the initiation of the intervention
  Drop-out and treatment retention

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik G Roozen, PhD, Principal Investigator — University of New Mexico; Department of Psychology/ CASAA
Locations (6):
- Netherlands (6):
  - IrisZorg, Arnhem, Gelderland
  - IrisZorg, Doetinchem, Gelderland
  - IrisZorg, Ede, Gelderland
  - IrisZorg, Nijmegen, Gelderland
  - IrisZorg, Tiel, Gelderland
  - IrisZorg, Zevenaar, Gelderland

IPD SHARING:
Plan to Share IPD: No